CLINICAL TRIAL: NCT03205436
Title: A Multi-center, Randomized Controlled Clinical Trial Evaluating the Effect of Fresh Amniotic Membrane in the Treatment of Diabetic Foot Ulcers: Crossover Group From Standard of Care
Brief Title: Affinity Prospective Diabetic Foot Trial Crossover Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organogenesis (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-DFU-AFF-02
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Graft (Experimental): Affinity human amniotic membrane
  Interventions: Other: Affinity human amniotic membrane

INTERVENTIONS:
Other: Affinity human amniotic membrane — fresh hypothermically stored human amniotic membrane

SUMMARY:
This study is an extension of the randomized controlled trial NT-DFU-AFF-01. Subjects that were randomized to the Standard of Care group will be able to crossover to the NT-DFU-AFF-02 trial and receive Affinity fHSAM if certain criteria are met.

DETAILED DESCRIPTION:
This study is an extension of the randomized controlled trial NT-DFU-AFF-01 in which subjects were randomized to SOC for 12 weeks or SOC and fresh hypothermically stored human amniotic membrane (Affinity; fHSAM) for 12 weeks to determine if addition of fHSAM to SOC results in faster healing of Wagner grade 1 and 2 DFUs compared to SOC alone.

At 6 weeks, patients from this RCT (NT-DFU-AFF-01) with study DFUs that have not been reduced in area by at least 40% will be exited from the study and considered treatment failures. This group (Group 2C) will constitute the active population in this single arm study (NT-DFU-AFF-02). Study wounds will receive up to 12 weeks of continuing SOC and fHSAM.

The standard of care therapy in this study is offloading of the DFU, appropriate sharp or surgical debridement, and aggressive infection management with the use of appropriate dressings (defined later in the protocol). A number of offloading systems are commercially available. The choice of offloading will be at the discretion of the principal investigator but should be total contact casting, fixed ankle walker boot, or equivalent device to the fixed ankle walker boot.

The Screening Phase (1 day) consists of a series of screening assessments designed to determine eligibility followed by, for those who meet the eligibility criteria (described in more detail below), treatment. At the Screening Visit (S1), written informed consent from the subject will be obtained by the Investigator or suitably qualified designee before the performance of any other protocol-specific procedure. The Screening Period is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study.

The Treatment Phase (12 Weeks) begins on the same day as the screening visit. During the Treatment Phase, subjects will be evaluated on a weekly basis. Efficacy evaluations each week will include Investigator assessment of ulcer healing and measurements of ulcer size using digital photographic planimetry. Safety evaluations during the Treatment Phase will consist of adverse event assessments at each visit.

Subjects whose ulcers do not achieve closure at 12 weeks or who experience an amputation will be deemed treatment failures.

ELIGIBILITY:
Inclusion Criteria:

1. A percentage area reduction of less than 40% after having received 6 weeks of treatment with SOC in the NT-DFU-01 trial.
2. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
3. Subject has read and signed the IRB/IEC approved Informed Consent Form.
4. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
5. At least 18 years old.

Exclusion Criteria:

1. Failure to complete 6 weeks of SOC in the original NT-DFU-01 study
2. Any AE or SAE that occurred during the NT-DFU-01 study, which, in the opinion of the investigator would preclude the subject successfully having Affinity applied for up to 12 weeks.
3. Subject is unlikely to complete a regimen of Affinity and SOC for up to 12 weeks due to personal reasons.
4. Subject is pregnant or breast feeding.
5. Osteomyelitis or bone infection of the affected foot as assessed by X-ray.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Time to initial closure of diabetic foot ulcer | 12 weeks

SECONDARY OUTCOMES:
Proportion of healed wounds | 12 weeks
Mean wastage of graft | 12 weeks
  healed wounds only
Mean cost to heal | 12 weeks
  healed wounds only

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - GF Professional Research, Miami Lakes, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - The Foot and Ankle Wellness Center, Ford City, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - SerenaGroup Research Institute, Pittsburgh, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No